CLINICAL TRIAL: NCT06450210
Title: Safety for Home Administration of Microdose Psilocybin Use
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Private Philanthropic Funds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: IRB00422973
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Psychedelic Experiences

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a double-blind study. Participants will be told they will receive a range of psilocybin doses (maximum 4.2 mg) and "at least one" dose of placebo. This will control for expectancy effects on cognitive testing and questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1.2 mg psilocybin trihydrate microdose (Experimental): Participants will receive a single microdose of 1.2 mg psilocybin trihydrate via oral capsule in the laboratory in double-blind fashion.
  Interventions: Drug: psilocybin trihydrate
- 2.0 mg psilocybin trihydrate microdose (Experimental): Participants will receive a single microdose of 2.0 mg psilocybin trihydrate via oral capsule in the laboratory in double-blind fashion.
  Interventions: Drug: psilocybin trihydrate
- 3.0 mg psilocybin trihydrate microdose (Experimental): Participants will receive a single microdose of 3.0 mg psilocybin trihydrate via oral capsule in the laboratory in double-blind fashion.
  Interventions: Drug: psilocybin trihydrate
- 4.2 mg psilocybin trihydrate microdose (Experimental): Participants will receive a single microdose of 4.2 mg psilocybin trihydrate via oral capsule in the laboratory in double-blind fashion.
  Interventions: Drug: psilocybin trihydrate
- Placebo (Placebo Comparator): Participants will receive a single placebo oral capsule in the laboratory in double-blind fashion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: psilocybin trihydrate — Microdoses of psilocybin trihydrate will be administered to participants (1.2 mg, 2.0 mg, 3.0 mg, and 4.2 mg).
  Arms: 1.2 mg psilocybin trihydrate microdose; 2.0 mg psilocybin trihydrate microdose; 3.0 mg psilocybin trihydrate microdose; 4.2 mg psilocybin trihydrate microdose
Drug: Placebo — Participants will receive a capsule identical in appearance to the active drug that contains an inactive substance.
  Arms: Placebo

SUMMARY:
The goal of this laboratory study is to establish whether and which microdoses of psilocybin are safe to administer at home to healthy participants.

Eligible participants will be given ascending doses of psilocybin trihydrate and a single, interspersed, randomized placebo on separate days in double-blind fashion. The participants will be asked to complete questionnaires and undergo safety assessments.

DETAILED DESCRIPTION:
This study aims to enroll 20 healthy participants who will complete all study procedures. Participants will undergo a standard screening procedure. Baseline measures will be completed before the first dose. Participants will then be given ascending doses of psilocybin trihydrate (1.2 mg, 2.0 mg, 3.0 mg, and 4.2 mg) and a single, interspersed, randomized placebo on separate days in double-blind fashion at the research site. A 1 mg dose of psilocybin anhydrate is equivalent to a 1.19 mg dose of psilocybin trihydrate (used in this study). For each session, participants will be assessed with criteria for the safety of home dosing. If any dose meets criteria for at-home dosing, and a lower dose did not fail these criteria, that dose will be identified as the safe dose for the given participant. After administration of all doses of psilocybin to all participants, if a safe at-home dose was identified for all participants, that will be considered the highest safe dose for at-home administration to be used for future studies.

Visit summary:

Initial screening: Medical and psychological screening (Approx. 4 hours though portions of this may be completed remotely).

Dosing sessions: There will be 5 double-blind laboratory dosing sessions involving administration of ascending doses of psilocybin and a single, interspersed, randomized placebo dose. Baseline questionnaires will be completed on the day of the first dosing visit, and safety assessments will be administered during and at the end of each session.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 60 years old
* Have given written informed consent
* Have at least a high-school level of education or equivalent (e.g. GED) and be fluent in English
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine.
* Agree not to take any as needed (PRN) medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Licensed to drive (for driving simulator test).

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g. atrial fibrillation, corrected QT interval (QTc) > 450 msec), artificial heart valve, or transient ischemic attack (TIA) in the past year
* Epilepsy
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive drugs (prescribed or not) on a daily basis. This includes nicotine but excepts caffeine.
* Currently taking on a regular (e.g. daily) basis any medications having a centrally-acting serotonergic effect, including monoamine oxidase inhibitors (MAOIs). For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least five half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table
* History of schizophrenia spectrum disorder
* History of bipolar I disorder
* History of substance induced psychotic disorder
* Current history of meeting Diagnostic and Statistical Manual (DSM)-5 criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine)
* Have a first degree relative with bipolar I disorder, or schizophrenia spectrum disorder.

Cardiovascular screening: To qualify for the study, blood pressure at screening will be less than 130 mmHg systolic, 80 mmHg diastolic, and 90 beats per minute; mean heart rate must also be no less than 40 beats per minute. Blood pressure will be taken while subjects are at rest and have been seated or supine for at least 5 minutes.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood pressure (mmHg) | Baseline, 1-4 hours post dose
  Blood pressure will be measured at 60, 120, 180, and 240 minutes. A dose will be deemed safe for home dosing if participants do not have elevations in blood pressure beyond threshold values; systolic blood pressure > 150 mmHg, diastolic blood pressure > 90mmHg) at any timepoint.
Heart rate in beats per minute (bpm) | Baseline; 1-4 hours post dose
  Heart rate will be measured at 60, 120, 180, and 240 minutes. A dose will be deemed safe for home dosing if participants do not have elevations in heart rate beyond threshold value of > 110 bpm
Field sobriety testing | Baseline; 90 minutes post dose
  The standardized battery of field sobriety tests includes: The Walk-and-Turn (W&T), One-Leg Stand (OLS), Horizontal Gaze Nystagmus (HGN). A dose will be deemed safe for home dosing if participants pass field sobriety testing at time of expected peak psilocybin effects.
  The cumulative amount of clues observed across these tasks (out of a possible 22 clues) will be reported.
Number of participants with normal or abnormal psychological status as assessed by a psychiatric mental status exam | 120 minutes post dose
  The Psychiatric Mental Status Exam will be a clinical interview identical to that performed by psychiatrists in daily clinical practice and will assess and document the participant's mood, affect, thought process (including the presence of formal thought disorder), paranoia, delusions, hallucinations, other perceptual alterations, speech (including rate, volume, prosody, whether or not speech is pressured), suicidal thoughts, and orientation to person, place and time. A dose will be deemed safe for home dosing if there is no evidence of abnormal psychological status on a psychiatric mental status exam performed by a blinded study psychiatrist.
  There is no formal scoring rubric for this outcome. A psychiatrist will use their clinical judgment to evaluate whether a participant has normal or abnormal psychological status based on a clinical interview.

SECONDARY OUTCOMES:
Driving Performance as assessed by The Systems Technology, Inc. Simulation (STISIM) Drive® M4000-R Console | Baseline; 60 minutes post dose
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. Specific driving outcomes include: lateral control (i.e., SDLP), longitudinal control (i.e., standard deviation of speed (SDSP), mean speed, number of speed exceedances), total accidents (sum of number of collisions, pedestrians hit, etc.), total rule violations (sum of number of missed stop signs, illegal turns, etc.), and distance to lead vehicles.
  Scores range from 0 to no upper limit. Higher scores represent higher magnitude of driving impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep M. Nayak, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- 5510 Nathan Shock Drive, Baltimore, Maryland, United States